CLINICAL TRIAL: NCT01379287
Title: A Phase I, Open-Label, Dose-Escalation Safety and Pharmacokinetic Study of Iso-Fludelone in Patients With Advanced Solid Tumors
Brief Title: Dose-Escalation Safety and Pharmacokinetic Study of Iso-Fludelone in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Pittsburgh (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-202
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumors
Keywords: Iso-Fludelone; KOS-1803; Dose-Escalation; 10-202

ARMS (1):
- Patients with Advanced Solid Tumors (Experimental): The trial was initially designed as a 3 hour IV infusion of iso-fludelone every 3 weeks with three dose-escalation stages (12 patients), however it has been amended to study iso-fludelone administered over 6 hours (+/- 30 minutes) every 3 weeks schedule.
  Interventions: Drug: Iso-Fludelone

INTERVENTIONS:
Drug: Iso-Fludelone — Iso-fludelone will be administered IV over 6 hours (+/- 30 mins) on Day 1 of every 3 week cycle.
  Other Names: KOS-1803

SUMMARY:
Iso-fludelone is a type of chemotherapy drug called an epothilone. Epothilones are drugs that attach to proteins in your body called "tubulins". Tubulins help cells to grow, and are found in both normal and cancer cells. When research animals with cancer were given the study drug, Iso-fludelone, the drug attached itself to "tubulin" and slowed or stopped the cancer cells from growing. Other types of epothilones have been tested in cancer patients and were found to be safe. A similar epothilone drug and other drugs called taxanes are currently approved by the FDA for treating certain types of cancers.

The purpose of this study is to see the effects, good and/or bad, of this investigational drug, Iso-fludelone, on cancer. The term "investigational" means the study drug being tested has not been approved by the United States Food and Drug Administration (FDA) or other regulatory agencies. This study is the first time the investigators are using iso-fludelone in people. This is a Phase I study. In a Phase I study, the first people to receive the drug are given a fairly low dose.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of malignancy at Memorial Sloan-Kettering Cancer Center
* Diagnosis of advanced stage, primary or metastatic adult solid tumors refractory to standard therapy or for which no curative standard therapy exists
* Evidence of radiographically measurable or non-measurable disease by RECIST 1.1 criteria.
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 4.0) Grade ≤1
* Age must be ≥ 18 years
* Last dose of antineoplastic therapy except for hormonal therapy must be > 21 days.
* Patients with brain metastasis that have been treated and clinically stable following intervention with neurological signs or symptoms resolved to CTCAEv4 Grade ≤1
* ECOG performance status must be 0 or 1.
* Required baseline laboratory data within 14 days of iso-fludelone administration include
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophils count ≥ 1.5 x 109 /L
* Platelet count ≥ 75 x 109 /L
* Serum bilirubin < or = to 1.5 x ULN
* AST and ALT < or = to 2.5 x ULN
* Serum creatinine < or = to 1.5 x ULN
* Willing and able to comply with scheduled visits, treatment plan, and laboratory tests.

Exclusion Criteria:

* Pre-existing diarrhea uncontrolled with supportive care. Prior hemorrhagic diarrhea due to ulcerative colitis, inflammatory bowel disease or other cause. Active, uncontrolled peptic ulcer disease (patients maintained with ranitidine or its equivalent are acceptable to enroll).
* Pre-existing neurological disease (including but not limited to peripheral sensory or motor neuropathy, seizures, gait disturbances, or tremors/involuntary movements) of CTCAEv4 Grade ≥ 2 due to any cause.
* Hypersensitivity reaction (CTCAEv4 Grade ≥ 2) to prior therapy containing hydroxypropyl-β-cyclodextrin, ethanol, propylene glycol, or patient may not be safely administered ethanol (e.g., current history of ethanol abuse or concomitant administration of Antabuse®).
* Concurrent therapy with any other investigational agent.
* Pregnant or breast-feeding women. Female patients must agree to use effective contraception, must be surgically sterile, or must be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate. All at-risk female patients must have a negative serum pregnancy test within 10 days prior to the start of study treatment.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV); prior myocarditis from any cause; pre-existing Grade 2 or higher arrhythmias ("non-urgent medical attention indicated").
* Dementia or altered mental status that would prohibit informed consent.
* Patients with untreated central nervous system (CNS) metastases.
* Patients with known leptomeningeal metastasis
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.
* Pre-existing ophthalmologic conditions (including glaucoma; history of demyelinating disease; vasculitis; retinal vascular occlusion and any optic neuropathy).
* History (or family history) of long QT syndrome or QTc > 450 msec on baseline ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2011-06-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | 2 years
  The MTD is defined as the dose that results in DLT in 25% of all evaluable patients.
To determine the dose limiting toxicity (DLT), safety | 2 years
  Toxicities and adverse events will be assessed using the NCI CTC version 4.0

SECONDARY OUTCOMES:
To evaluate the plasma pharmacokinetics of iso-fludelone when administered intravenously | over 6 hours (+/- 30 minutes) on a day 1 every 21 days schedule
  All PK analyses will be performed using the WinNonlin computer program; version 5.3 Pharsight Corporation, Mountain View, CA). PK Model selection will be based on a visual inspection of goodness of fit plots (observations vs. predictions, residuals and weighted residuals vs. predictions). The assay values (concentrations vs times) will be used to calculate individual-specific elimination rate constant (Ke), time to maximum Iso-fludelone concentration (Tmax), maximum Iso-fludelone concentration (Cmax) and area under the concentration-time curve (AUC) values.
To describe and assess any preliminary evidence of anti-tumor activity of iso-fludelone | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal Gounder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Christner SM, Parise RA, Levine ED, Rizvi NA, Gounder MM, Beumer JH. Quantitative method for the determination of iso-fludelone (KOS-1803) in human plasma by LC-MS/MS. J Pharm Biomed Anal. 2014 Nov;100:199-204. doi: 10.1016/j.jpba.2014.08.007. Epub 2014 Aug 12. PMID 25168219
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm